CLINICAL TRIAL: NCT00665457
Title: Neoadjuvant Therapy and Biomarker Analysis of Stage II and III Breast Cancer With Docetaxel/Capecitabine and Celecoxib Followed by Doxorubicin/Cyclophosphamide and Celecoxib
Brief Title: Biomarkers in Women Receiving Chemotherapy & Celecoxib for Stage II or Stage III Breast Cancer Removable by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study drug was removed from the market and low enrollment.
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0085-04-FB; P30CA036727 (NIH)
Record Dates: First submitted 2008-04-22; First posted 2008-04-23 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Capecitabine; Celecoxib; Cyclophosphamide; Docetaxel; Doxorubicin; liposomal doxorubicin; Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis; Reverse Transcriptase Polymerase Chain Reaction; Immunohistochemistry; Pharmacogenomic Testing; Biopsy, Needle; Neoadjuvant Therapy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Celecoxib (Experimental): •Neoadjuvant chemotherapy: Patients receive docetaxel IV over 1 hour on days 1, 8, and 15, oral capecitabine twice daily on days 1-14, and oral celecoxib twice daily on days 1-21. Courses repeat every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  Patients then receive doxorubicin hydrochloride IV and cyclophosphamide IV once daily on day 1, oral celecoxib twice daily on days 1-14, and filgrastim subcutaneously once daily on days 3-10. Courses repeat every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Celecoxib is stopped one week prior to surgery.
  •Surgery: Patients undergo definitive surgery (either modified radical mastectomy or lumpectomy combined with axillary node dissection). Patients may also undergo adjuvant radiotherapy and hormonal therapy at the discretion of multidisciplinary breast team.
  Interventions: Biological: filgrastim; Drug: capecitabine; Drug: celecoxib; Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin hydrochloride; Genetic: gene expression analysis; Genetic: polymorphism analysis; Genetic: protein expression analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: imaging biomarker analysis; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: pharmacogenomic studies; Procedure: dynamic contrast-enhanced magnetic resonance imaging; Procedure: needle biopsy; Procedure: neoadjuvant therapy; Procedure: radiomammography; Procedure: ultrasound imaging

INTERVENTIONS:
Biological: filgrastim
  Other Names: Neupogen
Drug: capecitabine
  Other Names: Xeloda
Drug: celecoxib
  Other Names: Celebrex
Drug: cyclophosphamide
  Other Names: Cytoxan, Neosar
Drug: docetaxel
  Other Names: Docefrez, Taxotere
Drug: doxorubicin hydrochloride
  Other Names: Lipodox, Lipodox 50, and Doxil
Genetic: gene expression analysis
Genetic: polymorphism analysis
Genetic: protein expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: imaging biomarker analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: pharmacogenomic studies
Procedure: dynamic contrast-enhanced magnetic resonance imaging
Procedure: needle biopsy
Procedure: neoadjuvant therapy
Procedure: radiomammography
Procedure: ultrasound imaging

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This phase II clinical trial is studying biomarkers and side effects in women receiving chemotherapy and celecoxib for stage II or stage III breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the safety and efficacy of four courses of neoadjuvant chemotherapy comprising docetaxel, capecitabine, and celecoxib followed by doxorubicin hydrochloride, cyclophosphamide, and celecoxib for the treatment of women with resectable stage II or III breast cancer.
* To determine the mRNA and protein levels of thyraidylate synthase (TS), thymidine phosphylase (TP), vascular endothelial growth factor (VEGF), Multi-Drug Resistance Protein 1 (MDR-1), cyclooxygenase-2 (COX-2), and matrix metalloproteinase-2 (MMP-2) in tumor tissue prior to and following treatment.
* To correlate baseline expression of TS, TP, VEGF, MDR, COX-2, and MMP-2 to tumor response measured by physical exam, breast MRI, breast ultrasound, mammography, and pathologic response.
* To determine if polymorphisms in the genes that encode those proteins also correlate with outcome, if a correlation is found between specific molecular markers and clinical outcome.

OUTLINE:

* Neoadjuvant chemotherapy: Patients receive docetaxel IV over 1 hour on days 1, 8, and 15, oral capecitabine twice daily on days 1-14, and oral celecoxib twice daily on days 1-21. Courses repeat every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients then receive doxorubicin hydrochloride IV and cyclophosphamide IV once daily on day 1, oral celecoxib twice daily on days 1-14, and filgrastim subcutaneously once daily on days 3-10. Courses repeat every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Celecoxib is stopped one week prior to surgery.

* Surgery: Patients undergo definitive surgery (either modified radical mastectomy or lumpectomy combined with axillary node dissection). Patients may also undergo adjuvant radiotherapy and hormonal therapy at the discretion of multidisciplinary breast team.

Blood is collected at baseline and examined for genetic polymorphisms associated with functional changes in proteins. Tumor tissue is obtained by needle biopsy at baseline, before the second course of docetaxel/capecitabine/celecoxib, and at surgical resection. Molecular markers and protein expression are assessed by immunohistochemistry using fluorescence-image analysis and real-time reverse-transcriptase PCR.

Patients undergo imaging comprising dynamic MRI, ultrasound, and mammogram at baseline and after the first and second 4 courses of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic evidence of invasive breast cancer

  * Stage II-III disease
  * Resectable disease
* Must have a primary tumor estimated by mammogram, ultrasound or palpation to be ≥ 3 cm and/or palpable axillary nodes > 1 cm for whom neoadjuvant chemotherapy is appropriate
* ECOG performance status 0-1
* Absolute granulocyte count > 2,000/mm^3
* Platelet count > 100,000/mm^3
* Serum bilirubin < 1.5 times upper limit of normal (ULN)
* Serum creatinine < 1.5 times ULN
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* At least 2 weeks since prior treatment with cyclooxygenase (COX)-2 inhibitors

Exclusion Criteria:

* Not pregnant or nursing/negative pregnancy test
* No allergies to sulfa medication, aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs)
* No uncontrolled concurrent illness that might jeopardize the patient's ability to receive the chemotherapy program outlined in this protocol, including any of the following:

  * Active infection requiring intravenous antibiotics
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Serious, uncontrolled cardiac arrhythmia
* No other prior malignancy except for adequately treated basal cell or squamous cell skin cancer, noninvasive carcinomas, or other cancers from which the patient has been disease-free for at least 5 years
* No prior chemotherapy or radiation therapy for ipsilateral breast cancer
* No concurrent sorivudine or brivudine to treat herpes simplex or herpes zoster viral infections
* No concurrent participation in another therapeutic clinical trial

Ages: 19 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-04-15 (Actual); Primary Completion 2009-07-31 (Actual); Study Completion 2009-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C. Reed, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Celecoxib: •Neoadjuvant chemotherapy: Patients receive docetaxel IV over 1 hour on days 1, 8, and 15, oral capecitabine twice daily on days 1-14, and oral celecoxib twice daily on days 1-21. Courses repeat every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  Patients then receive doxorubicin hydrochloride IV and cyclophosphamide IV once daily on day 1, oral celecoxib twice daily on days 1-14, and filgrastim subcutaneously once daily on days 3-10. Courses repeat every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Celecoxib is stopped one week prior to surgery.
  •Surgery: standard of care
Period: Overall Study
Arm/Group | Celecoxib
Started | 3
Completed (All three subjects completed chemotherapy treatment and went on to surgery.) | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Celecoxib
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 46.3 [40 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 4 Adverse Events
Description: Grading of adverse events was determine by the principal investigator according to NCI common toxicity criteria (CTC version 3.0). Safety analysis is based on any participant experiencing a grade 4 AE.
Time Frame: every 3 weeks X 4, then every 2 weeks X4
Population: Of the 3 participants, one had a grade 4 event - neutropenic fever.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 3
Participants | 1

2. Primary Outcome: Participants Who Experienced Pathologic Complete Response, Progression-free and Overall Survival, and Time to Treatment Failure
Description: CTEP RECIST guidelines are defined as followed: Pathologic complete response is no signs of residual malignancy cells at the primary site and axillary lymph nodes are seen with histologic examination. Progression-free survival is defined as from the first date of therapy until the first notation of clinical progression or relapse. Overall survival is defined as from the first date of therapy until the date of death. Time to treatment failure is defined as from the first date of therapy until the date the patient is removed from study for any reason.
Time Frame: 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 3
Participants
  pathologic complete response | 0
  progression free survival | 1
  overall survival | 1
  time to treatment failure | 1

ADVERSE EVENTS:
Arm/Group | Celecoxib
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib (N=3)
Neutropenic Fever (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=3)
Weight Loss (Metabolism and nutrition disorders) | 1
Paronychia (Immune system disorders) | 3
Elevated Liver Enzymes (Hepatobiliary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Lacrimal Stenosis (Eye disorders) | 2
Intractable nausea and vomiting (Gastrointestinal disorders) | 1
Neutropenic fever (Immune system disorders) | 1
Obstruction nasolacrimal duct (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No